CLINICAL TRIAL: NCT05447260
Title: A New Prognostic Stratification-based Safety and Efficacy Study of Ruxolitinib in Myelofibrosis: a Multicenter, Prospective, Single-arm Clinical Study
Brief Title: A New Prognostic Stratification-based Safety and Efficacy Study of Ruxolitinib in Myelofibrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIPSS70+2.0 MF
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ruxolitinib (Experimental)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Dosage based on platelet count

SUMMARY:
This is a multi-center, prospective, single-arm study to assess safety and efficacy of Ruxolitinib in myelofibrosis (MF) based on a new prognostic stratification.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years with a diagnosis of primary or secondary MF by World Health Organization and International Working Group for Myeloproliferative Neoplasms Research and Treat- ment (IWG-MRT) criteria;
2. Received ruxolitinib treatment for ≥3 months.

Exclusion Criteria:

1. Malignant tumors with other progression or myelofibrosis secondary to other diseases;
2. Exclude myelofibrosis patients after splenectomy;
3. Patients with poor compliance with case follow-up or lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a ≥35% reduction in palpable spleen volume from baseline. | From Week 0 through Week 24
  Reduction in spleen volume is measured by magnetic resonance imaging/computerized tomography (MRI/CT).

SECONDARY OUTCOMES:
The proportion of patients with ≥50% reduction in Total Symptom Score (TSS) from baseline. | From Week 0 through Week 24
  TSS is assessed by the MPN-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided